CLINICAL TRIAL: NCT05176860
Title: Evaluation of Novel Cone-Beam CT for Guidance and Adaptation of Precision Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAR-2021-12
Record Dates: First submitted 2021-12-16; First posted 2022-01-04 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer; Liver Cancer; Breast Cancer; Other Cancer
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-site study designed to generate data describing the quality and applicability of on-couch high-performance CBCT imaging for anatomy visualization and radiation treatment dosimetry planning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- High-performance CBCT imaging (Experimental): Two additional study imaging sets are acquired.
  Interventions: Device: CBCT Imaging

INTERVENTIONS:
Device: CBCT Imaging — Two research CBCT images will be acquired per subject.

SUMMARY:
This is a feasibility study investigating the image quality of a new, high-performance cone beam CT (CBCT) used for on-couch imaging during radiotherapy treatments.

DETAILED DESCRIPTION:
This study focuses on potential benefits of a high performance cone beam CT (CBCT) image guidance system for improved precision in the delivery of radiotherapy. CBCT is currently used during radiation therapy to align the patient to their original treatment plan to increase the precision of radiation delivery. Current CBCT imaging technology requires approximately a minute to acquire an image. In order to acquire images with sufficient quality to allow accurate targeting, the patient may need to perform multiple breath hold maneuvers to "freeze" the motion of tumors that move with the breathing cycle (e.g. lung, liver, and breast tumors). The new high-performance CBCT can acquire an image in approximately 6 seconds, potentially enabling acquisition of images with a single breath hold. Improved motion compensation algorithms used in image reconstruction may allow acquisition of good quality images even while a patient is not holding their breath.

The methodology for the subject's treatment setup, CT simulation, treatment planning, image guidance and treatment delivery will be determined by the subject's treatment team and is not specified by this study. Enrollment in the study may occur after treatment delivery has started but must be prior to the fifth fraction.

Following completion of informed consent to participate in this study, high-performance CBCT imaging will be scheduled immediately before or after one of the subject's first five scheduled radiation treatment fractions. Two research CBCT images will be acquired, one with breath hold, the other with free breathing.

With minimal disruption for participating patients, this study will enable a comparison of (i) the subject's treatment planning fan-beam CT and (ii) the conventional CBCT acquired on an existing treatment unit with (iii) the high-performance CBCT. Image quality of the high performance CBCT image data will thereby be compared to both a best-case standard (fan-beam) and the status-quo for on-couch imaging to isolate and identify improvements.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for treatment on one of the five TrueBeam platforms at the NS Health QE2 site.
* Subject is receiving radiation therapy using a breath-hold technique (for example, lung, liver and left breast cancers).

Exclusion Criteria:

* Patient is pregnant or has plans for pregnancy during the period of treatment.
* Patient is unwilling to consent to participating to the study, or for whom informed consent is not possible.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
CBCT Image Quality | 1 day
  The quality of fan-beam CT, standard CBCT and high-performance CBCT will be evaluated by calculating contrast, noise, resolution, Hounsfield Unit accuracy and artifact reduction.
  Furthermore, the three image sets will be evaluated qualitatively by multiple observers with training in radiation oncology and image-guided radiation therapy, who will rank the images acquired for each subject by perceived quality/usefulness for structure contouring and RT guidance.

SECONDARY OUTCOMES:
Dosimetry Calculations | 1 day
  Dose-volume histograms for key target structures and organs at risk will be calculated from both the high-performance and standard CBCT images and compared to those from the existing dosimetric plan for each subject to determine the accuracy of the dosimetric calculations based on the CBCTs.
Patient Experience | 1 day
  The patient experience with CBCT image acquisition will be determined through the use of a questionnaire comparing elements of the standard CBCT image acquisition process to that of the high-performance CBCT process.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health (QEII), Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No